CLINICAL TRIAL: NCT06711510
Title: Predict to Prevent PGRN Disease
Acronym: PREVENT-PGRN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: loss of funding
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240482
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Frontotemporal Dementia (FTD); GRN Related Frontotemporal Dementia
Keywords: Frontotemporal dementia; frontotemporal lobar degeneration; GRN; PGRN; mutation; , neurofilament light chain (NfL); biomarker; amyotrophic lateral sclerosis; primary progressive aphasia
MeSH Terms: conditions — Frontotemporal Dementia; Frontotemporal Lobar Degeneration; Charcot-Marie-Tooth disease, Type 1F; Amyotrophic Lateral Sclerosis; Aphasia, Primary Progressive | interventions — Blood Specimen Collection; Spinal Puncture

STUDY DESIGN:
Intervention Model Description: Nine evaluations (every 3 months) over a 2-year follow-up, with the same standardized protocol for all participants, including:
  * At the inclusion visit (M0), after 12 months (M12) and after 24 months (M24):
    * clinical (neurological) evaluation
    * behavioral examination
    * cognitive testing
    * blood sampling (determination of carrier / non-carrier status by means of GRN testing will be done at M0 visit; results will remain strictly confidential and not disclosed to study participants and investigators)
    * brain MRI
    * olfactory swab sampling with nasal brush
    * skin punch biopsy (optional)
    * lumbar puncture for CSF sampling (optional)
  * For the remaining visits (M3, M6, M9, M15, M18, M21):
    * clinical evaluation
    * blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standardized protocol for all participants (Other): Nine evaluations (every 3 months) over a 2-year follow-up, with the same standardized protocol for all participants, including:
  * At the inclusion visit (M0), after 12 months (M12) and after 24 months (M24):
    * clinical (neurological) evaluation
    * behavioral examination
    * cognitive testing
    * blood sampling (determination of carrier / non-carrier status by means of GRN testing will be done at M0 visit; results will remain strictly confidential and not disclosed to study participants and investigators)
    * brain MRI
    * olfactory swab sampling with nasal brush
    * skin punch biopsy (optional)
    * lumbar puncture for CSF sampling (optional)
  * For the remaining visits (M3, M6, M9, M15, M18, M21):
    * clinical evaluation
    * blood sampling
  Interventions: Other: Clinical, behavioral and cognitive evaluation; Other: blood sampling; Other: brain MRI; Other: olfactory swab sampling with nasal brush; Other: skin punch biopsy; Other: lumbar puncture for CSF sampling

INTERVENTIONS:
Other: Clinical, behavioral and cognitive evaluation — Questionnaries and tests
Other: blood sampling — blood sampling (56ml max)
Other: brain MRI — brain MRI (35 to 70 minutes)
Other: olfactory swab sampling with nasal brush — olfactory swab sampling with nasal brush
Other: skin punch biopsy — skin punch biopsy (optional intervention)
Other: lumbar puncture for CSF sampling — lumbar puncture for CSF sampling (optional intervention)

SUMMARY:
Progranulin (GRN or PGRN) mutations are among the most common genetic causes of frontotemporal lobar degeneration (FTLD). With the advent of gene-specific therapeutic interventions, an accurate knowledge of the presymptomatic phase of the disease is of utmost importance. Increases of plasma neurofilament light chain (NfL) levels are good predictors of phenoconversion in presymptomatic carriers. However their increase rates remain partially elucidated insofar, with many confounding factors. Another point which deserves further precision is the definition of the biological onset of the disease, via the identification of markers of intraneuronal accumulation of TDP-43 protein. PREVENT-PGRN aims aims at studying the trajectory of plasma NfL changes in presymptomatic GRN mutation carriers in comparison with healthy controls, in partnership with the GENFI-QBS study. Additionally, other disease-related biomarkers, namely associated with TDP-43 pathology, will be investigated in this study, at the presymptomatic and clinical phase.

DETAILED DESCRIPTION:
Despite several advances in the understanding of the presymptomatic phase of GRN-associated FTLD, some aspects concerning longitudinal biomarker changes and their capacity to predict phenoconversion have been only partially elucidated. Plasma NfL levels proved to be good tools for monitoring neurodegeneration in the years preceding phenoconversion, but thresholds for cross-sectional values and longitudinal increase rates need to be validated in international studies on large populations. In addition, numerous confounding factors (head trauma, epilepsy, metabolic disorders, etc.) may punctually impact plasma NfL dosages. This may suggest that several measurements spaced over time are best predictors of phenoconversion rather than a single assay. Whether cross-sectional NfL levels or their rate of change during follow-up are the best parameter for individual monitoring in the presymptomatic and clinical phases still has to be determined. This knowledge is an essential prerequisite for all current and future therapeutic trials designed for GRN carriers at the presymptomatic phase.

To answer this question, this project aims to define the trajectory of plasma NfL levels as exactly as possible in carriers of GRN gene mutations during the presymptomatic and clinical phase. NfL dosages will be performed every 3 months over a 2-year period and carriers' trajectories will be compared with those measured in age-matched control individuals. This study takes place in the frame of the international collaborative project GENFI-QBS substudy (quarterly blood sampling), aiming at characterizing the evolution of plasma biomarkers in genetic FTLD by repeated assays every 3 months. Plasma samples will also allow complementary biomarker analyses, providing a broader biomarker panel to better elucidate the pathophysiological mechanisms of the disease. Notably, the validation of in vivo TDP-43 biomarkers and the tracking of the longitudinal progression of the proteinopathy represent other major challenges. Indeed, the advent of such a biomarker in asymptomatic GRN carriers would allow to establish the start of the lesional process (i.e., TDP-43 accumulation) and thus the appropriate moment to start preventive treatments.

Therefore, this study will enrol 90 participants, including 10 patients with early-stage FTD (or other clinically defined syndromes within FTLD spectrum) carrying pathogenic GRN mutations and 80 asymptomatic at-risk individuals (i.e., first-degree relatives of individuals carrying a GRN mutation. These latter will thus be either presymptomatic GRN carriers (~50% risk) or controls. The determination of the genetic status of asymptomatic participants will be done in research setting, and results will be blinded to participants and investigators. A part of study participants will be selected from Predict-PGRN (NCT04014673), a natural history study aiming at characterizing the presymptomatic phase of PGRN disease over 5-year follow-up.

A comprehensive evaluation including neurological examination, cognitive and behavioral assessment, brain MRI, biological blood sampling and olfactory swab sampling will be performed at inclusion, at 12 months and at 24 months. Neuropsychological, behavioral and MRI data will allow to compare additional cognitive-behavioral and neuroimaging markers between carriers and non-carriers, providing further information on the clinical progression and the risk of phenoconversion of the former. As optional assays, upon participants' specific consent, CSF sampling and skin biopsy will be proposed at the same time-points, in order to provide additional substrates to look for biomarkers of TDP-43 accumulation, together with plasma and olfactory mucosa samples. Intermediate visits will be made every 3 months (at month 3, 6, 9, 15, 18 and 21), only for quick clinical follow-up and blood sampling. The purpose of these visits is to enable close monitoring of blood biomarkers, namely NfL, but also to document the occurrence of intercurrent events and to monitor participants' clinical status.

ELIGIBILITY:
Inclusion Criteria:

* For all :

  * signature of informed consent for the study
  * being French speaker
  * having social security coverage
  * absence of any other neurological disease
* For asymptomatic at-risk individuals :

  * being first-degree relative of a GRN mutation carrier OR of a patient suffering from FTD with discovery of a GRN mutation in their family
  * absence of any neurological troubles related to the disease
* For patients :

  * being carrier of a pathogenic GRN mutation
  * diagnosis of behavioural-variant frontotemporal dementia according to Rasckvsky et al. criteria (2011) or any related clinical syndromes, such as primary progressive aphasia according to Gorno-Tempini et al. criteria (2011)

Exclusion Criteria:

* For all :

  * any contraindication to brain MRI (pace-maker, ferromagnetic heart valve, aneurysm clips or any other ferromagnetic foreign body implanted in brain/eye or other critical locations, non-MRI compatible intrauterine devices, claustrophobia)
  * chronic alcohol use / addiction
  * known chronic kidney disease
  * hypersensitivity to local anaesthetics
  * impossibility of laying down for 1 hour without moving
  * pregnant of breastfeeding women, or any beta-HCG positive test for women in childbearing age N.B.: participation in therapeutic essays is not an exclusion criteria, but should be discussed with the study investigator in every case.
* For asymptomatic at-risk individuals :

  * Peaple under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Compare the trajectory of plasma NfL between GRN mutation carriers, during the presymptomatic and clinical phases, and non-carrier controls, to improve identification of early disease phases and guide future therapeutic trials. | 2 years
  Cross-sectional and longitudinal comparisons of NfL assays by Simoa® technique on plasma samples collected every 3 months during the 9 study visits (M0, M3, M6, M9, M12, M15, M18, M21, M24), between GRN mutation carriers and non-carrier controls.

SECONDARY OUTCOMES:
Compare the levels of other known biomarkers of interest in fluids (plasma, CSF) (such as GFAP, for example) between GRN mutation carriers, during the presymptomatic and clinical phases, and non-carrier controls. | 2 years
  Cross-sectional comparisons of other fluid biomarkers known to be associated with FTLD disease (e.g., GFAP) sampled every 3 months for 2 years (9 time-points) between GRN mutation carriers and controls.
Compare the trajectory of other known biomarkers of interest in fluids (plasma, CSF) mentioned above (such as GFAP, for example) between carriers of GRN gene mutations, during the presymptomatic and clinical phases, and non-carrier controls. | 2 years
  Longitudinal comparisons of the trajectories of other fluid biomarkers known to be associated with FTLD disease (e.g., GFAP) sampled every 3 months for 2 years (9 time-points) between GRN mutation carriers and controls.
Discover new fluid biomarkers (plasma, CSF) and peripheral biomarkers (nasal mucosa, fibroblasts) targeting, in particular, the detection of the TDP-43 protein (by RT-QuIC, among others). | 2 years
  Comparisons of the level of new fluid (plasma, CSF) and peripheral (nasal brush, skin biopsy) biomarkers targeting TDP-43 pathology between patients, presymptomatic carriers and controls.
Establish correlations between biomarker trajectories and neuropsychological profiles | 2 years
  Correlations between the levels of measured biomarkers with neuropsychological and behavioral scores obtained at each yearly visit (3 time-points).
Establish correlations between biomarker trajectories and neuroimaging profiles | 2 years
  Correlations between the levels of measured biomarkers with structural and functional neuroimaging data obtained at each yearly visit (3 time-points).

IPD SHARING:
Plan to Share IPD: No